CLINICAL TRIAL: NCT05084534
Title: Efficacy and Safety of Midodrine in Refractory or Recurrent Ascites in Children With Cirrhosis - A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Midodrine in Refractory or Recurrent Ascites in Children With Cirrhosis.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No cases of refractory ascites presented to hospital in one year
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-47
Record Dates: First submitted 2021-10-18; First posted 2021-10-19 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2021-10

CONDITIONS: Refractory Ascites in Children With Cirrhosis
MeSH Terms: interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midodrine hydrochloride plus standard medical treatment (Experimental): * Standard Medical Treatment will be continued in all, which includes,
  * To continue restriction of sodium to < 2meq/kg/day
  * To continue maximum tolerable dose of diuretics
  * Repeat LVP with infusion of albumin (8 g/L) performed for tense, symptomatic ascites
  * Albumin infusion for serum albumin <2.5g/dl - dose 1g/kg/day (maximum 20g/day)
  * Midodrine starting at 0.25mg/kg/day in divided doses, increased to 0.5mg/kg/day after 7 days if MAP does not increase by >10% (maximum dose - 15mg/day)
  * Midodrine dosage will be decreased by 25% in case of arterial hypertension (>95th centile BP for the age)
  Interventions: Drug: Midodrine; Other: Standard medical treatment
- Standard medical treatment (Other): * Standard Medical Treatment will be continued in all, which includes,
  * To continue restriction of sodium to < 2meq/kg/day
  * To continue maximum tolerable dose of diuretics
  * Repeat LVP with infusion of albumin (8 g/L) performed for tense, symptomatic ascites
  * Albumin infusion for serum albumin <2.5g/dl - dose 1g/kg/day (maximum 20g/day)
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: Midodrine — Midodrine starting at 0.25mg/kg/day in divided doses, increased to 0.5mg/kg/day after 7 days if MAP does not increase by >10% (maximum dose - 15mg/day)
  • Midodrine dosage will be decreased by 25% in case of arterial hypertension (>95th centile BP for the age)
  Arms: Midodrine hydrochloride plus standard medical treatment
Other: Standard medical treatment — Standard Medical Treatment will be continued in all, which includes,
  * To continue restriction of sodium to < 2meq/kg/day
  * To continue maximum tolerable dose of diuretics
  * Repeat LVP with infusion of albumin (8 g/L) performed for tense, symptomatic ascites
  * Albumin infusion for serum albumin <2.5g/dl - dose 1g/kg/day (maximum 20g/day)

SUMMARY:
Refractory ascites is seen in 17% of cirrhotic patients with the 1year mortality rate being high, upto 20-50% [1]. The pathogenesis of cirrhotic ascites includes release of vasodilatory molecules like nitric oxide, damage associated molecular pathogens (DAMPs) and pattern associated molecular pathogens (PAMPs) secondary to bacterial translocation, which causes splanchnic bed vasodilation resulting in activation of renin-angiotensin and aldosterone axis causing sodium and water retention. The standard medical therapy for the treatment of ascites includes sodium restriction to 2mEq/kg/day with diuretics (Spirinolactone 3-6mg/kg/day and furosemide 0.5-2 mg/kg/day) and therapeutic paracentesis (>50ml/kg/day) with albumin replacement at 8g/L of ascitic fluid tapped. Refractory ascites is defined as ascites that cannot be mobilized by sodium - restricted diet (maximum upto 2mEq/kg/day- 88meq=2gm of salt) and high-dose diuretic treatment (6 mg/kg/day of spironolactone and 2 mg/kg/day of furosemide) or optimum doses of diuretics cannot be given due to development of diuretic-induced complications (Sodium <130mEq, AKI as per KDIGO, hypovolemia, hypo (<3.5meq)/hyperkalemia (>5meq); new onset HE) and recurrent ascites as ascites that has recurred within a 12 weeks period despite standard treatment. All the children and adolescents upto 18 years of age with refractory or recurrent ascites will be included in the study and randomized into 2 groups. One group will receive only standard medical therapy and other group will receive midodrine and standard medical therapy for 12 weeks. Mean arterial pressure will be monitored at every OPD visit. At the end of 12 weeks, plasma renin activity, number of therapeutic paracentesis done, change in serum sodium, estimated glomerular filtration rate and complications will be assessed.

If there is complete resolution of ascites, liver transplantation or death before 12 weeks, midodrine will be stopped.

DETAILED DESCRIPTION:
Aim: To determine the efficacy of midodrine in combination with standard medical therapy in reduction of refractory or recurrent ascites in children with cirrhosis

Primary objective:

• To compare the proportion of patients who will achieve partial or complete control of ascites at 12 weeks after therapy between the two groups

Secondary Objectives:

* Comparison of total number of therapeutic paracentesis (>50ml/kg) procedures between the groups by the end of 12 weeks
* Frequency of complete response (elimination of ascites) by 12 weeks
* Time taken to achieve complete response
* Frequency of partial response (persistent ascites not requiring therapeutic paracentesis) by 12 weeks
* To compare change in plasma renin activity from baseline to 12 weeks
* Change in serum sodium from baseline to 4 weeks and 12 weeks
* Change in eGFR from baseline to 4 weeks
* Change in MAP at 1 week, 4 weeks and 12 weeks from baseline
* Comparison of proportion of patients with transplant free survival at 12 weeks between the 2 groups
* Frequency of worsening HE by 12 weeks
* Frequency of development of HRS by 12 weeks
* Proportion of patients developing hypertension at 12 weeks
* Frequency of development of adverse effects by 12 weeks

Methodology:

* Study population : Children and Adolescents with cirrhosis and refractory or recurrent ascites with stable renal function (age appropriate creatinine level in last 2 weeks) attending the Pediatric Hepatology Department
* Study design:

Open label RCT (computer based randomization - block randomization with block size of 4)

* Study period:12 weeks for each patient; The study will be conducted between September 2021 and December 2022
* Sample size: Pilot study - 10 patients in each group

  * Intervention:
  * Standard Medical Treatment will be continued in all, which includes,
  * To continue restriction of sodium to < 2meq/kg/day
  * To continue maximum tolerable dose of diuretics
  * Repeat LVP with infusion of albumin (8 g/L) performed for tense, symptomatic ascites
  * Albumin infusion for serum albumin <2.5g/dl - dose 1g/kg/day (maximum 20g/day)
  * Midodrine starting at 0.25mg/kg/day in divided doses, increased to 0.5mg/kg/day after 7 days if MAP does not increase by >10% (maximum dose - 15mg/day)
  * Midodrine dosage will be decreased by 25% in case of arterial hypertension (>95th centile BP for the age)

Monitoring and assessment :

* Abdominal girth, Blood pressure (MAP) , HE - every visit (1-2 weekly)
* Haemogram, INR, Liver function test, Kidney function test- every 2 weekly
* Bedside Ultrasound - every visit (1-2 weekly)
* Plasma renin activity at baseline and 12 weeks
* Need for therapeutic paracentesis (tense ascites causing respiratory embarrassment) at every visit (1-2 weekly)

Adverse effects: Hypertension , Bradycardia, Piloerection, Pruritus, Dysuria

Stopping rule of the study:

* Complete resolution of ascites or 12 weeks of midodrine therapy whichever is earlier
* Liver transplantation
* Death without transplantation
* TIPSS

ELIGIBILITY:
Inclusion Criteria:

* • Children and Adolescents of age group upto 18 years with cirrhosis and refractory Ascites that cannot be mobilized by sodium - restricted diet (maximum upto 2mEq/kg/day- 88meq=2gm of salt) and high-dose diuretic treatment (6 mg/kg/day of spironolactone and 2 mg/kg/day of furosemide) or optimum doses of diuretics cannot be given due to development of diuretic-induced complications (Sodium <130mEq, AKI as per KDIGO, hypovolemia, hypokalemia (<3.5meq)/hyperkalemia (>5meq); new onset HE) or ascites that recurs within 4 weeks of mobilization) or recurrent ascites ( Ascites that has recurred 3 times within 12 months despite standard medical treatment) with stable renal function (age appropriate creatinine level in last 2 weeks) attending the Pediatric Hepatology Department, ILBS will be prospectively included in this study after informed consent.

Exclusion Criteria:

1. GIT bleeding in last 1 month
2. SBP in last 1 month
3. HE grade 3 or higher
4. Septic shock
5. Hepatorenal syndrome
6. Presence of PVT
7. Renal or cardiovascular disease or arterial hypertension
8. Presence of HCC

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
• To compare the proportion of patients who will achieve partial or complete control of ascites at 12 weeks after therapy between the two groups | 12 weeks

SECONDARY OUTCOMES:
• Comparison of total number of therapeutic paracentesis (>50ml/kg) procedures between the groups by the end of 12 weeks | 12 weeks
• Frequency of complete response (elimination of ascites) by 12 weeks | 12 weeks
• Time taken to achieve complete response | 12 weeks
• Frequency of partial response (persistent ascites not requiring therapeutic paracentesis) by 12 weeks | 12 weeks
• To compare change in plasma renin activity from baseline to 12 weeks | 12 weeks
• Change in serum sodium from baseline to 4 weeks and 12 weeks | 12 weeks
• Change in eGFR from baseline to 4 weeks | 4 weeks
• Change in MAP at 1 week, 4 weeks and 12 weeks from baseline | 12 weeks
• Comparison of proportion of patients with transplant free survival at 12 weeks between the 2 groups | 12 weeks
• Frequency of worsening HE by 12 weeks | 12 weeks
• Frequency of development of HRS by 12 weeks | 12 weeks
• Proportion of patients developing hypertension at 12 weeks | 12 weeks
• Frequency of development of adverse effects by 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ILBS, New Delhi, India